CLINICAL TRIAL: NCT05004142
Title: Evaluation of the Antitumor Activity, Safety, and Pharmacokinetic Profile of FCN-437c in Combination With Fulvestrant or Letrozole + Goserelin in Female Patients With ER+, HER2- Advanced Breast Cancer
Brief Title: Study of Efficacy, Safety, and Pharmacokinetics of FCN-437c in Combination With Fulvestrant or Letrozole+Goserelin
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahon Pharmaceutical Co., Ltd. (Other)
Collaborators: Hebei Medical University Fourth Hospital (Other); The First Hospital of Jilin University (Other); Affiliated Hospital of Hebei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AH150202-1
Record Dates: First submitted 2021-06-15; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-06

CONDITIONS: Breast Neoplasms
Keywords: ER-Positive; HER2-Negative; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FCN-437c with Fulvestrant (Experimental): FCN-437c 200mg, oral administration under fasting conditions, QD, for 21 days, with 7-day discontinuation, 28 days for 1 cycle; Fulvestrant, C1D1 and C1D15 and Day 1 of each cycle, 500mg/day, intramuscularly.
  Interventions: Drug: FCN-437c+Fulvestrant
- FCN-437c in combination with Letrozole + Goserelin (Experimental): FCN-437c 200mg, oral administration under fasting conditions, QD, for 21 days, with 7-day discontinuation, 28 days for 1 cycle; Letrozole 2.5 mg, QD, for continuous dosing; Goserelin 3.6 mg, subcutaneously, once every 28 days.
  Interventions: Drug: FCN-437c+Letrozole+Goserelin

INTERVENTIONS:
Drug: FCN-437c+Fulvestrant — FCN-437c 200mg, oral administration under fasting conditions, QD, for 21 days, with 7-day discontinuation, 28 days for 1 cycle; Fulvestrant, C1D1 and C1D15 and Day 1 of each cycle, 500mg/day, intramuscularly.
  Arms: FCN-437c with Fulvestrant
Drug: FCN-437c+Letrozole+Goserelin — FCN-437c 200mg, oral administration under fasting conditions, QD, for 21 days, with 7-day discontinuation, 28 days for 1 cycle; Letrozole 2.5 mg, QD, for continuous dosing; Goserelin 3.6 mg, subcutaneously, once every 28 days.
  Arms: FCN-437c in combination with Letrozole + Goserelin

SUMMARY:
This is a multicenter, open-label clinical study to evaluate the safety and antitumor activity of FCN-437c in combination with Fulvestrant for the treatment of post-menopausal female patients with ER+ and HER2- advanced breast cancer, FCN-437c in combination with Letrozole + Goserelin for the treatment of pre-menopausal female patients with ER+ and HER2- advanced breast cancer, and to evaluate the PK characteristics of the FCN-437c combination therapies.

This study is consist of two cohorts, Cohort 1: FCN-437c in combination with Fulvestrant (1st or 2nd line treatment for postmenopausal ER+, HER2-advanced breast cancer); Cohort 2: FCN-437c in combination with Letrozole + Goserelin (1st line treatment for premenopausal ER+, HER2- advanced breast cancer). Thirty patients will be enrolled in each cohort, for a total of 60 patients.

Tumor Assessment:

Tumor evaluation will be performed every 8 weeks (±7 days) according to RECIST version 1.1 until disease progression, withdrawal of informed consent, or death; for patients who discontinue the drug due to toxicity, imaging evaluation is required until disease progression.

End of Treatment and End of Study:

End of Study (EOS) is defined as 2 years after the last patient's first dose or the end of treatment (whichever is earlier). At the end of the study, the investigator will decide whether the patients whose disease has not progressed shall continue taking FCN-437c and other combination agents or not based on clinical benefit.

Cohort 1: Post-menopausal patients diagnosed with ER+, HER2- advanced breast cancer, who have not received prior systemic therapy for advanced breast cancer, or who have disease progression determined by imaging assessment during their 1st line endocrine therapy; Cohort 2: Pre-menopausal patients diagnosed with ER+, HER2- advanced breast cancer, who have not received prior systemic therapy for advanced breast cancer;

DETAILED DESCRIPTION:
Screening period (Day-28 to Day-1);

* Continuous dose treatment period: 28 days for each treatment cycle, with patients evaluated every 8 weeks until disease progression, withdrawal of informed consent or death; for patients discontinued due to toxicity, imaging evaluation is required until disease progression;
* Follow-up after the end of treatment (within 30 days from the last dose);
* Survival follow-up (once telephone follow-up every 3 months until the end of study);

Primary Objectives:

* To observe the efficacy and safety of continuous oral administration of FCN-437c in combination with Fulvestrant in post-menopausal female patients with ER+, HER2- advanced breast cancer;
* To observe the efficacy and safety of continuous oral administration of FCN-437c in combination with Letrozole + Goserelin in pre-menopausal female patients with ER+, HER2- advanced breast cancer;

Secondary Objectives:

* To characterize the PK profile of FCN-437c in combination with Letrozole + Goserelin;
* To characterize the PK profile of FCN-437c in combination with Fulvestrant; End of study: 2 years after the last patient's first dose or the end of treatment (whichever is earlier);

ELIGIBILITY:
Inclusion Criteria:

* Subjects are eligible to be included in the study only if they meet all of the following criteria:

  1. Patients with advanced breast cancer diagnosed as ER+, HER2-; ER+ is defined as histologically or cytologically confirmed ER+ with positive nuclear staining of estrogen receptor tumor cells ≥ 1% by immunohistochemistry; HER2- is defined as histologically or cytologically confirmed HER2-, with a negative ISH test result or an IHC test result of 0, 1+, or 2+, and if the IHC test result is 2+, the ISH test result must be negative;
  2. Criteria of menopausal status and prior treatment, and see Appendix 3 for definition of menopause:

     Cohort 1 (FCN-437c in combination with Fulvestrant): post-menopausal patients with advanced breast cancer, who are not suitable for curative surgical resection or radiation therapy and have not previously received systemic therapy, or have disease progression supported by imaging evaluation during their first-line endocrine therapy (including anti-estrogen or aromatase inhibitors).

     Cohort 2 (FCN-437c in combination with Letrozole + Goserelin): pre-menopausal patients with advanced breast cancer, who are not suitable for curative surgical resection or radiation therapy and have not received systemic therapy; Note: If any relapse or metastases occur within 12 months from the treatment start during the (neo) adjuvant endocrine therapy or within 12 months after the (neo) adjuvant endocrine therapy, such (neo) adjuvant endocrine therapy will be taken as one line of systemic therapy.
  3. ECOG (Eastern Cooperative Oncology Group) performance status score at 0 or 1;
  4. According to RECIST 1.1, patients must have at least one measurable lesion ( for any lesion received radiotherapy or other local treatments, it may be considered as a measurable lesion if disease progression is proved by radiographic evidence after completion of treatment).

     Note: Patients with only bone metastases must have at least one bone lesion that is predominantly osteolytic if no measurable lesion is present (for patients with no measurable lesion and only one osteolytic lesion, if prior radiotherapy to that lesion was performed, it is eligible if radiographic evidence supports disease progression of this bone lesion after radiotherapy).
  5. Life expectancy for at least 12 weeks;
  6. The bone marrow and organ function of the patient should be adequate:

     1. Absolute neutrophil count ≥1.5×109/L;
     2. Hemoglobin ≥ 90 g/L (without erythrocyte transfusion in 14 days);
     3. Platelets ≥75×109/L;
     4. Serum total bilirubin ≤1.5×ULN (upper limit normal), and ≤3.0×ULN for patients with Gilbert's syndrome;
     5. AST (aspartate aminotransferase), ALT(alanine aminotransferase) ≤2.5×ULN; for patients with liver metastasis, both AST and ALT should be ≤5×ULN;
     6. Creatinine < 1.5×ULN and creatinine clearance ≥50mL/min (Ccr=((140-age) × body weight (kg))/(72×Scr (mg/dl)) or Ccr=((140-age) × body weight (kg))/(0.818×Scr (umol/L)) Note: For females, the results should be calculated by × 0.85).
  7. Willingness and ability to comply with planned visits, treatment plans, laboratory tests and other trial procedures;
  8. Subject should fully understand this study and agree to sign the ICF (informed consent form).

Exclusion Criteria:

* Patients that meet any of the following conditions shall not be included in this clinical study:

  1. Prior treatment criteria:

     1. Prior treatment with a CDK4/6 inhibitor;
     2. Prior systemic chemotherapy for advanced breast cancer;
     3. Prior radiotherapy, major surgery, immunotherapy, monoclonal antibody therapy and other systemic anti-tumor therapy within 4 weeks before initiation of study drug administration;
     4. Cohort 1:

     i. (a) Previously received two or more lines of endocrine therapy; If relapse or metastases occur within 12 months from the treatment start during the (neo) adjuvant endocrine therapy or within 12 months after the (neo) adjuvant endocrine therapy, such (neo) adjuvant endocrine therapy will be taken as one line of systemic therapy; ii. Previously received Fulvestrant as first-line endocrine therapy for advanced breast cancer; e) Cohort 2: i. Previously treated with systemic anti-tumor therapy including endocrine therapy for advanced breast cancer; Note: Patients with disease progression after more than 12 months from the initiation or completion of the (neo) adjuvant therapy are eligible; Patients received Tamoxifen or an aromatase inhibitor within 14 days or an LHRH analogue within 28 days are eligible.
  2. Patients unsuitable for endocrine therapy due to metastases to any important organ or with large tumor loads, e.g., patients judged by the investigator to be unsuitable for endocrine therapy:

     1. symptomatic visceral metastases;
     2. rapid disease progression or impaired visceral functions;
     3. Non-visceral metastases requiring chemotherapy based on the investigator's clinical judgment;
  3. Failure to recover from toxic effects of prior anti-tumor therapy (> grade 2 as defined by NCI-CTCAE version 5.0);
  4. Receipt strong CYP3A inhibitors (amprenavir, atazanavir, boceprevir, clarithromycin, conivaptan, delavirdine, diltiazem, erythromycin, fosamprenavir, indinavir, itraconazole, ketoconazole, lopinavir, mibefradil, miconazole, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin, verapamil, voriconazole, etc.) or strong CYP3A inducers (carbamazepine, felbamate, nevirapine, phenobarbital, phenytoin, primidone, rifabutin, rifampin, rifapentine, etc.) within 14 days before the first dose;
  5. Cardiac function and diseases that meet one of the following conditions:

     1. 12-lead electrocardiogram (ECG) measurements at the study site during the screening period, with a QTcF > 470 ms based on the QTcF formula;
     2. Arrhythmia with clinical significance, including but not limited to complete left bundle branch block and second-degree atrioventricular block;
     3. Any risk factors prolonging the QTc interval, such as hypokalemia, inherited long QT syndrome, use of drugs that prolong the QTc interval (mainly including Class Ia, Class Ic and Class III antiarrhythmic drugs; for drugs potentially prolong the QTc interval, see https://crediblemeds.org/index.php/tools/pdfdownload? f=cql_en; e.g., haloperidol, droperidolum, chloroquine, quinidine, procainamide, disopyramide, sotalol, amiodarone, doxepin, mianserin, mexiletine, loratadine, etc.).
     4. Cardiac failure congestive with New York Heart Association (NYHA) classification ≥ Class 3;
  6. Difficulty in swallowing, or with an active digestive disorder, or with major GI surgery, or with malabsorption syndrome, or other conditions that may impair the absorption of FCN-437c (e.g., ulcerative lesions, uncontrollable nausea, vomiting, diarrhea, malabsorption syndrome, and small bowel resection).
  7. Known hypersensitivity to the study drugs Letrozole, Fulvestrant, Goserelin, or to FCN-437c or any excipients;
  8. Uncontrolled CNS metastases, unless all of the following requirements are met:

     1. More than 4 weeks after radiotherapy or surgery before the start of the study treatment;
     2. CNS metastases are clinically stable, asymptomatic and do not require hormonal or other dehydration therapy;
     3. No meningeal metastases;
  9. Active infection, including patients with positive hepatitis B surface antigen (HBsAg), and HBV DNA ≥1.00×103 IU/ml; patients with positive hepatitis C virus antibody (Anti-HCV); patients infected with human immunodeficiency virus (HIV);
  10. For Cohort 2 only:

      i. Pregnant or lactating women; ii. For female patients of childbearing potential, disagreeing to use an effective contraceptive method, such as double barrier methods, condoms and or IUDs, during treatment and for at least 30 days after the last dose of the study treatment;
  11. Any other diseases or conditions with clinical significance that investigators believe may affect the compliance with the protocol or patients' signature of ICF, such as uncontrollable diabetes, active or uncontrollable infections;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — A Multicenter, Open-label Phase II Clinical Study: Evaluation of the Antitumor Activity, Safety, and Pharmacokinetic Profile of FCN-437c in Combination with Fulvestrant or Letrozole + Goserelin in female patients with ER+, HER2- Advanced Breast Cancer
Enrollment: 70 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | through study completion, assessed up to 24 months
  Overall response rate (ORR) of FCN-437c in combination of fulvestrant in post-menopausal patients and letrozole + goserelin in pre-menopausal patients based on RECIST 1.1

SECONDARY OUTCOMES:
Safety and tolerability of the combination therapy | Up to 30 days after EOT
  Assessed by grade and frequency of adverse events, serious adverse events, AEs leading to permanent drug discontinuation and death and changes in lab values, vital signs, ECGs, physical examinations and ECOG status.
PFS | through study completion, assessed up to 24 months
  Progression free survival (PFS) during the treatment.
OS | through study completion, assessed up to 24 months
  overall survival (OS) during the treatment.
1-year overall survival rate | through study completion, assessed up to 24 months
  1-year OS rate during the treatment.
DOR | through study completion, assessed up to 24 months
  duration of response (DOR) during the treatment.
CBR | through study completion, assessed up to 24 months
  Clinical benefit response (CBR) during the treatment.
PK parameters of FCN-437c combination therapy Cmax | Plasma concentration of FCN-437c and PK parameters
  Plasma concentration of FCN-437c and PK parameters
PK parameters of FCN-437c combination therapy AUC | Plasma concentration of FCN-437c and PK parameters
  Plasma concentration of FCN-437c and PK parameters
PK parameters of FCN-437c combination therapy Tmax | Plasma concentration of FCN-437c and PK parameters
  Plasma concentration of FCN-437c and PK parameters

CONTACTS AND LOCATIONS:
Overall Officials: Yunjiang Liu, Doctor, Principal Investigator — Hebei Medical University Fourth Hospital
Locations (1):
- Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slamon DJ, Neven P, Chia S, Fasching PA, De Laurentiis M, Im SA, Petrakova K, Bianchi GV, Esteva FJ, Martin M, Nusch A, Sonke GS, De la Cruz-Merino L, Beck JT, Pivot X, Vidam G, Wang Y, Rodriguez Lorenc K, Miller M, Taran T, Jerusalem G. Phase III Randomized Study of Ribociclib and Fulvestrant in Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Advanced Breast Cancer: MONALEESA-3. J Clin Oncol. 2018 Aug 20;36(24):2465-2472. doi: 10.1200/JCO.2018.78.9909. Epub 2018 Jun 3. PMID 29860922
- [Background] Im SA, Lu YS, Bardia A, Harbeck N, Colleoni M, Franke F, Chow L, Sohn J, Lee KS, Campos-Gomez S, Villanueva-Vazquez R, Jung KH, Chakravartty A, Hughes G, Gounaris I, Rodriguez-Lorenc K, Taran T, Hurvitz S, Tripathy D. Overall Survival with Ribociclib plus Endocrine Therapy in Breast Cancer. N Engl J Med. 2019 Jul 25;381(4):307-316. doi: 10.1056/NEJMoa1903765. Epub 2019 Jun 4. PMID 31166679
- [Background] Sledge GW Jr, Toi M, Neven P, Sohn J, Inoue K, Pivot X, Burdaeva O, Okera M, Masuda N, Kaufman PA, Koh H, Grischke EM, Frenzel M, Lin Y, Barriga S, Smith IC, Bourayou N, Llombart-Cussac A. MONARCH 2: Abemaciclib in Combination With Fulvestrant in Women With HR+/HER2- Advanced Breast Cancer Who Had Progressed While Receiving Endocrine Therapy. J Clin Oncol. 2017 Sep 1;35(25):2875-2884. doi: 10.1200/JCO.2017.73.7585. Epub 2017 Jun 3. PMID 28580882
- [Background] Cristofanilli M, Turner NC, Bondarenko I, Ro J, Im SA, Masuda N, Colleoni M, DeMichele A, Loi S, Verma S, Iwata H, Harbeck N, Zhang K, Theall KP, Jiang Y, Bartlett CH, Koehler M, Slamon D. Fulvestrant plus palbociclib versus fulvestrant plus placebo for treatment of hormone-receptor-positive, HER2-negative metastatic breast cancer that progressed on previous endocrine therapy (PALOMA-3): final analysis of the multicentre, double-blind, phase 3 randomised controlled trial. Lancet Oncol. 2016 Apr;17(4):425-439. doi: 10.1016/S1470-2045(15)00613-0. Epub 2016 Mar 3. PMID 26947331
- See also: Phase III Randomized Study of Ribociclib and Fulvestrant in Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Advanced Breast Cancer: MONALEESA-3 — https://pubmed.ncbi.nlm.nih.gov/?term=Im+SA&cauthor_id=29860922
- See also: Overall Survival with Ribociclib plus Fulvestrant in Advanced Breast Cancer — https://pubmed.ncbi.nlm.nih.gov/31826360/
- See also: Ribociclib plus endocrine therapy for premenopausal women with hormone-receptor-positive, advanced breast cancer (MONALEESA-7): a randomised phase 3 trial — https://pubmed.ncbi.nlm.nih.gov/29804902/
- See also: Overall Survival with Ribociclib plus Endocrine Therapy in Breast Cancer S.-A. Im, Y.-S. Lu, A. Bardia, N. Harbeck, M. Colleoni, F. Franke, L. Chow, J. Sohn, K.-S. Lee, S. Campos-Gomez, R. Villanueva-Vazquez, K.-H. Jung, A. Chakravartty, G. Hughes, I. — https://pubmed.ncbi.nlm.nih.gov/31166679/
- See also: MONARCH 2: Abemaciclib in Combination With Fulvestrant in Women With HR+/HER2- Advanced Breast Cancer Who Had Progressed While Receiving Endocrine Therapy — https://pubmed.ncbi.nlm.nih.gov/28580882/
- See also: hormone-receptor-positive, HER2-negative metastatic breast cancer that progressed on previous endocrine therapy (PALOMA-3) — https://pubmed.ncbi.nlm.nih.gov/26947331/
- See also: Overall Survival with Palbociclib and Fulvestrant in Advanced Breast Cancer — https://pubmed.ncbi.nlm.nih.gov/30345905/
- See also: The Effect of Abemaciclib Plus Fulvestrant on Overall Survival in Hormone Receptor-Positive, ERBB2-Negative Breast Cancer That Progressed on Endocrine Therapy-MONARCH 2: A Randomized Clinical Trial — https://pubmed.ncbi.nlm.nih.gov/31563959/